CLINICAL TRIAL: NCT02828462
Title: Impact of a Monitoring Device for Patients With Cancer Treated Using Oral Therapeutics
Acronym: CAPRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-A00254-47; 2016/2371 (Other: CSET Number)
Record Dates: First submitted 2016-06-29; First posted 2016-07-11 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Metastatic Cancer; Hematological Malignancy
MeSH Terms: conditions — Neoplasm Metastasis; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental: Patients using the device
  Interventions: Other: CAPRI
- Control: Patients not using the device

INTERVENTIONS:
Other: CAPRI
  Groups: Experimental

SUMMARY:
The emergence of oral delivery in cancer therapeutics is expected to result in an increased need for better coordination between all treatment stakeholders, mainly to ensure adequate treatment delivery to the patient. There is significant interest in the nurse navigation program's potential to improve transitions of care by improving communication between treatment stakeholders and by providing personalized organizational assistance to patients. The use of health information technology is another strategy aimed at improving cancer care coordination that can be combined with the NN program to improve remote patient follow-up. However, the potential of these two strategies combined to improve oral treatment delivery is limited by a lack of rigorous evidence of actual impact.

The investigators are conducting a large scale randomized controlled trial designed to assess the impact of a navigation program denoted CAPRI that is based on two Nurse Navigators and a web portal ensuring coordination between community and hospital as well as between patients and navigators, versus routine delivery of oral anticancer therapy. The primary research aim is to assess the impact of the program on treatment delivery for patients with metastatic cancer, as measured by Relative Dose Intensity. The trial involves a number of other outcomes, including toxic side effects, patient quality of life and patient experience . An economic evaluation adopting a societal perspective will be conducted, in order to estimate those health care resources' used. A parallel process evaluation will be conducted to describe implementation of the intervention

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female) aged > 18 years
* Life expectancy > 6 months
* Patients with tumour or hematological malignancy being treated at Gustave Roussy
* Patients with oral therapy (cytotoxic or targeted therapies)
* Patients starting therapy
* Patients living in France
* Patients affiliated to a social security system or equivalent
* OMS score from 0 to 2 at the time of inclusion
* Signed inform consent
* Patients able to follow protocol

Exclusion Criteria:

* Patients being treated with hormonotherapy only
* Patients enrolled in a clinical trial ongoing treatment with an experimental compound except in the case where the sponsor agrees that the CAPRI protocol is not intefering with the trial
* Not French speaking patients
* Patients deprived of liberty
* Patients with no internet access or telephone line

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic cancer or hematological malignancy being treated with oral therapy
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-10-24 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Relative dose intensity | Assessed every 30 days from randomization up to 6 months
  RDI will be calculated as follow "delivered dose intensity/dose intensity of the standard tumor regimen"

SECONDARY OUTCOMES:
Compliance | Assessed every 30 days from randomization up to 6 months
  Compliance will be assessed using Morisky questionnaire
Toxicity | Assessed every 30 days from randomization up to 6 months
  Grade 3 or 4 using NCICTCAE version 4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

REFERENCES:
- [Derived] Minvielle E, Perez-Torrents J, Salma I, Aegerter P, Ferrua M, Ferte C, Leleu H, Mathivon D, Sicotte C, Di Palma M, Scotte F. The Effect of Nurse Navigators in Digital Remote Monitoring in Cancer Care: Case Study Using Structural Equation Modeling. J Med Internet Res. 2025 Mar 28;27:e66275. doi: 10.2196/66275. PMID 40153795
- [Derived] Mir O, Ferrua M, Fourcade A, Mathivon D, Duflot-Boukobza A, Dumont S, Baudin E, Delaloge S, Malka D, Albiges L, Pautier P, Robert C, Planchard D, de Botton S, Scotte F, Lemare F, Abbas M, Guillet M, Puglisi V, Di Palma M, Minvielle E. Digital remote monitoring plus usual care versus usual care in patients treated with oral anticancer agents: the randomized phase 3 CAPRI trial. Nat Med. 2022 Jun;28(6):1224-1231. doi: 10.1038/s41591-022-01788-1. Epub 2022 Apr 25. PMID 35469070
- [Derived] Gerves-Pinquie C, Daumas-Yatim F, Lalloue B, Girault A, Ferrua M, Fourcade A, Lemare F, Dipalma M, Minvielle E. Impacts of a navigation program based on health information technology for patients receiving oral anticancer therapy: the CAPRI randomized controlled trial. BMC Health Serv Res. 2017 Feb 13;17(1):133. doi: 10.1186/s12913-017-2066-x. PMID 28193214